CLINICAL TRIAL: NCT01163253
Title: A Phase 3, Multi-Site, Open-Label Study Of The Long Term Safety And Tolerability Of 2 Oral Doses Of CP-690,550 In Subjects With Moderate To Severe Chronic Plaque Psoriasis
Brief Title: A Long Term Study To Evaluate The Safety And Tolerability Of CP-690,550 For Patients With Moderate To Severe Chronic Plaque Psoriasis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3921061; 2010-020002-15 (EudraCT Number)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis
Keywords: chronic; severe; treatment; safety; CP-690,55; Plaque Psoriasis; Psoriasis Vulgaris; Xeljanz; Tofacitinib
MeSH Terms: conditions — Psoriasis; Bronchiolitis Obliterans Syndrome; Lymphoma, Follicular | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Active Treatment (Experimental): The study is anticipated to continue for up to at least 2 years post First Market Approval (FMA) in a global, major market.
  All subjects will receive 10 mg BID of CP-690,550 for first 3 months of trial. Study has the option for variable dosing with 5 mg or 10 mg BID after first 3-months of treatment based on PI discretion
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — 5 mg oral BID
Drug: CP-690,550 — 10 mg oral BID

SUMMARY:
The main objective of this study is to evaluate the long-term safety of CP-690,550 in patients being treated for moderate to severe chronic plaque psoriasis. This is an open label extension study available to patients who participated in one of the qualifying studies with CP-690,550 providing entry criteria is met.

DETAILED DESCRIPTION:
The study terminated on 08MAR2016 as it met its objectives of characterizing long term safety and tolerability. The study did not terminate due to safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Have participated in qualifying study with CP-690,550 and are 18 years or older with diagnosis of plaque-type psoriasis (psoriasis vulgaris).

Exclusion Criteria:

* Non-plaque or drug induced forms of psoriasis;
* Cannot discontinue current oral, injectable or topical therapy for psoriasis or cannot discontinue phototherapy (PUVA or UVB).
* Any uncontrolled significant medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2867 (Actual)
Dates: Start 2010-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (320):
- United States (99):
  - Radiant Research, Inc., Birmingham, Alabama
  - UAB Dermatology, Birmingham, Alabama
  - Horizon Research Group, Inc., Mobile, Alabama
  - Radiant Research, Inc., Tucson, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Associates In Research, Inc., Fresno, California
  - University of California Irvine, Irvine, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists, Inc., Oceanside, California
  - MedDerm Associates, San Diego, California
  - UCSD Dermatology, San Diego, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Clinical Science Institute, Santa Monica, California
  - Healthcare Partners Medical Group, Torrance, California
  - Cherry Creek Research, Inc., Denver, Colorado
  - The Savin Center, P.C., New Haven, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Florida Academic Dermatology Center, Coral Gables, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - International Dermatology Research, Inc., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Leavitt Medical Associates of Florida dba Ameriderm Research, Ormond Beach, Florida
  - Miami Research Associates, Inc., South Miami, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Atlanta Dermatology, Vein & Research Center, P.C., Alpharetta, Georgia
  - Advanced Medical Research, Inc., Atlanta, Georgia
  - MedaPhase Inc., Newnan, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Schaumburg Dermatology, Schaumburg, Illinois
  - NorthShore University Health System - Division of Dermatology, Skokie, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Dundee Dermatology, West Dundee, Illinois
  - Deaconess Clinic Downtown Research Institute, Evansville, Indiana
  - Hudson Dermatology, Evansville, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DermResearch, PLLC, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital - Clinical Unit for Research Trials and Outcomes in Skin, Boston, Massachusetts
  - Michigan Center for Research Corporation dba Michigan Center for Skin Care Research, Clinton, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre - Dermcenter, Troy, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Saint Louis University - Department of Dermatology, St Louis, Missouri
  - Skin Specialists, P.C, Omaha, Nebraska
  - Bettencourt Skin Center, Henderson, Nevada
  - Dartmouth-Hitchcock Medical Center-Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Centennial Center-Comprehensive Clinical Research, Berlin, New Jersey
  - New York University (NYU) School of Medicine - Investigational Pharmacy (IP Shipment, Pharmacy), New York, New York
  - NYU Langone Medical Center, Ambulatory Care Center, Department of Dermatology, Clinical Studies Unit, New York, New York
  - The Rockefeller University, New York, New York
  - University of North Carolina at Chapel Hill- Hospital, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Dermatology Consulting Services, High Point, North Carolina
  - Wake Dermatology Associates, LLC, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Dermatology Associates, Wilmington, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Piedmont Imaging, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Triad Dermatology, PA, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Jewish Hospital, Cincinnati, Ohio
  - Radiant Research, Inc., Cincinnati, Ohio
  - IP ONLY: University Hospitals Case Medical Center, Cleveland, Ohio
  - University Hospitals Case Medical Center/Dept. of Dermatology, Cleveland, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Baker Allergy Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center - Department of Dermatology, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Office of John Michael Humeniuk, MD, Greer, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Rivergate Dermatology Clinical Research Center, PLLC, Goodlettsville, Tennessee
  - Dermatology Associates of Knoxville PC, Knoxville, Tennessee
  - Dermatology Research Associates, Nashville, Tennessee
  - Arlington Research Center, Inc., Arlington, Texas
  - Dermatology Treatment & Research Center, Dallas, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates, PA, Houston, Texas
  - Office of Mark Lee, MD, San Antonio, Texas
  - Progressive Clinical research, P.A., San Antonio, Texas
  - Stephen Miller, MD, PA, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Rockwood Research Center, Spokane, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Mountain State Clinical Research, Bridgeport, West Virginia
  - Madison Skin and Research, Inc., Madison, Wisconsin
- Argentina (2):
  - Centro De Investigaciones Dermatologicas, Caba
  - CENIT Centro de Neurociencias Investigacion y Tratamiento, CABA
- Australia (5):
  - Dr. Glenn and Partners, Kogarah, New South Wales
  - Premier Dermatology, Kogarah, New South Wales
  - Malvern Diagnostic Imaging, Malvern, Victoria
  - Emeritus Research, Malvern East, Victoria
  - Skin And Cancer Foundation, Melbourne, Victoria
- Austria (2):
  - LKH Feldkirch, Feldkirch
  - LKH Salzburg, Landesklinik fuer Dermatologie, Salzburg
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- UHC Sarajevo, Sarajevo, Bosnia and Herzegovina
- Brazil (3):
  - Hospital da Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Instituto de Dermatologia e Estetica do Brasil LTDA - IDERJ, Rio de Janeiro
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Bulgaria (6):
  - UMHAT "Dr Georgi Stranski", Pleven
  - UMHAT "Dr. Georgi Stranski" - II clinical base, Pleven
  - Tsentar za kozhno venericheski zaboliavania EOOD, Sofia
  - Mnogoprofilna Bolnitsa Za Aktivno Lechenie- Tokuda Bolnitsa, Sofia
  - UMBAL-Alexandrovska- Sofia Klinika po dermatologia i venerologia, Sofia
  - MBAL na Voennomeditsinska Akademia, Sofia
- Canada (34):
  - Kirk Barber Research, Calgary, Alberta
  - Northwest Dermatology & Laser Centre, Calgary, Alberta
  - Stratica Medical, Edmonton, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Derm Research @888 Inc, Vancouver, British Columbia
  - The Skin Centre, Vancouver, British Columbia
  - Percuro Clinical Research Limited, Victoria, British Columbia
  - Dermadvances Research, Winnipeg, Manitoba
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Dr. Zohair Tomi PMC Inc. Paton Medical Centre, St. John's, Newfoundland and Labrador
  - NewLab Clinical Research Inc., St. John's, Newfoundland and Labrador
  - Eastern Canada Cutaneous Research Associates Ltd., Halifax, Nova Scotia
  - CCA Medical Research, Ajax, Ontario
  - The Waterside Clinic, Barrie, Ontario
  - Ultranova Skincare, Barrie, Ontario
  - Co-Medica Research Network Inc., Courtice, Ontario
  - Dermatrials Research, Inc., Hamilton, Ontario
  - The Guenther Dermatology Research Centre, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Oakville Dermatology Laser Centre, Oakville, Ontario
  - Dr. Tuppal's Privat Practice, Oshawa Clinic, Oshawa, Ontario
  - Office of Dr. Michael Robern, Ottawa, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Office of Dr. Paul Adam (back-up location), Scarborough Village, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Windsor Clinical Research, Windsor, Ontario
  - Innovaderm Research Inc, Montreal, Quebec
  - Siena Medical Research, Montreal, Quebec
  - CRCMRGilbert Inc., Centre de Dermatologie Maizerets, Québec, Quebec
  - Centre de Recherche Dermatologique du Québec Métropolitain, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Chile (3):
  - Clinica Dermacross S.A., Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos, CIEC, Santiago, Santiago Metropolitan
- Colombia (6):
  - Reumalab S.A.S., Medellín, Antioquia
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Centro Integral de Reumatologia del Caribe Cicaribe S.A.S, Barranquilla, Atlántico
  - Riesgo De Fractura S.A, Bogota, Cundinamarca
  - Colegio Mayor de Nuestra Señora del Rosario, Bogotá, Cundinamarca
  - Medicity S.A.S, Bucaramanga, Santander Department
- Croatia (3):
  - University Hospital Center Osijek, Osijek
  - University hospital center "Sestre milosrdnice" clinic for dermatology and venerology disease, Zagreb
  - University hospital center zagreb, Zagreb
- Czechia (8):
  - Nemocnice Ceske Budejovice, a.s. Ustavni lekarna, České Budějovice, Czech Republic
  - Ustanvi lekarna, Hradec Králové, Czech Republic
  - Nemocnice Ceske Budejovice,a.s., České Budějovice
  - Klinika nemoci koznich a pohlavnich, Hradec Králové
  - Fakultni nemocnice Plzen, Plzen-Bory
  - Kozni ordinace, Prague
  - Lekarna U sv. Ignace, Prague
  - Krajska zdravotni a.s.,Masarykovy nemocnice o.z., Ústí nad Labem
- Denmark (5):
  - Aarhus University Hospital, Aarhus C
  - Bispebjerg Hospital, University of Copenhagen, Copenhagen NV
  - Gentofte Hospital, Hellerup
  - Hudklinikken Herning, Herning
  - Hudklinikken, Svendborg
- Tampere Univeristy Hospital, Department of Dermatology and Venereology, Tampere, Finland
- France (17):
  - Chu Morvan, Brest, Cedex
  - CHU Limoges - Hôpital Dupuytren - Pharmacie, Limoges, Cedex
  - Hopital Saint Louis, Paris, Lle-de-france
  - Hôpital Jean Minjoz, Besançon
  - CHU Jean-Minjoz, Besançon
  - CHG Le Mans, Le Mans
  - Hopital Dupuytren, Limoges
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU De Nice Hopital De L'Archet II, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Lyon Sud - Pharmacie, Pierre-Bénite
  - C.H.U. de Poitiers la Miletrie, Poitiers
  - C.H.U de Reims, Reims
  - Hôpital Robert Debre, Reims
  - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Larrey Departement de Dermatologie, Toulouse
  - Hopital de Brabois / Batiment Philippe Canton, Vandœuvre-lès-Nancy
- Germany (29):
  - Universitaets-Hautklinik Eberhard-Karls-Universitaet Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Charité Universitätsmedizin Berlin, Berlin
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Facharzt fuer Dermatologie und Allergologie, Berlin
  - MVZ Reichenberger Str., Aerztehaus "Rudolf Virchow", Berlin
  - Hautarztpraxis Tegel, Berlin
  - Klinik and Poliklinik fur Dermatologie and Allergologie der Universitaet Bonn, Bonn
  - Klinik und Poliklinik fur Dermatologie und Allergologie der Universitaet Bonn, Bonn
  - Dres. Kirsten Prepeneit und Volker Streit, Buchholz
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinik Carl Gustav Carus, Dresden
  - Universitaetsklinikum Erlangen Hautklinik im Internistischen Zentrum, Erlangen
  - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt am Main
  - Universitaetsklinik und Poliklinik fuer Dermatologie und Venerologie, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Gemeinschaftspraxis Dres.Michael Ockenfels und Christoph Sauter, Hanau
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck, Lübeck
  - Hautarztpraxis Dres. Scholz, Sebastian, Schilling, Mahlow
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KoeR, Mainz
  - Technischen Universitaet Muenchen, München
  - Universitaetsklinikum Muenster, Münster
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Eberhard-Karls-Universitaet Tuebingen Universitaetshautklinik, Tübingen
  - HSK, Dr. Horst Schmidt Kliniken GmbH, Wiesbaden
  - Hautarztpraxis Centrovital, Witten
- Greece (3):
  - University Dermatology Clinic "Andreas Syggros" Hospital, Athens, Attica
  - University General Hospital of Ioannina / Dermatology and Venereology Department, Ioannina
  - "Papageorgiou" General Hospital/B' Dermatology and Venereology Clinic of University of Thessaloniki, Thessaloniki
- The University of Hong Kong (HKU)-Queen Mary Hospital (QMH), Hong Kong, Hong Kong
- Hungary (12):
  - Synexus Magyarorszag Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Borgyogyaszati Klinika, Debrecen
  - Bacs-Kiskun Megyei Korhaz Szegedi Tudomanyegyetem AOK Oktato Korhaza, Borgyogyaszati Osztaly, Kecskemét
  - Miskolci Semmelweis Korhaz es Egyetemi Oktatokorhaz, Borgyogyaszati Osztaly, Miskolc
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Klinikai Kutatasi Osztaly, Nyíregyháza
  - Szabolcs-Szatmar-Bereg Megyei Korjazak es Egyetemi Okatokorhaz, Borgyogyaszati Szakrendeles, Nyíregyháza
  - Pecsi Tudomanyegyetem Aok Bor- Nemikortani Es Onkodermatologiai Klinika, Pécs
  - SZTE Szentgyorgyi Albert Klinikai Kozpont/Borgyogyaszati es Allergologiai Klinika, Szeged
  - Tolna Megyei Balassa Janos Korhaz, Borgyogyaszati Osztaly, Szekszárd
  - ALLERGO-DERM BAKOS Kft., Szolnok
  - Vas Megyei Markusovszky Korhaz/Borgyogyaszati Osztaly, Szombathely
  - Veszprem Megyei Csolnoky Ferenc Korhaz Borgyogyaszat, Veszprém
- Japan (5):
  - Gunma University Hospital, Maebashi, Gunma
  - JR Sapporo hospital, Sapporo, Hokkaido
  - Kobe University, Kobe, Hyōgo
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
- Mexico (4):
  - Instituto Dermatologico De Jalisco "Dr Jose Barba Rubio", Zapopan, Jalisco
  - Mexico Centre for Clinical Research S.A. de C.V., Mexico City, Mexico City
  - Centro de Dermatologia de Monterrey, Monterrey, Nuevo León
  - Centro Medico San Lucas, Monterrey, Nuevo León
- Netherlands (2):
  - Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam, North Holland
  - PT&R, Beek
- Poland (16):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - NZOZ Zdrowie Osteo-Medic, Bialystok
  - Klinika Dermatologii, Wenerologii i Alergologii Uniwersyteckiego Centrum Klinicznego, Gdansk
  - Krakowskie Centrum Medyczne NZOZ, Krakow
  - Specjalistyczne Gabinety Lekarskie "Dermed", Lodz
  - Novum Instytut Dermatologii Leczniczej i Estetycznej, Opole
  - Solumed Centrum Medyczne, Poznan
  - Centrum Badan Klinicznych s.c. Wieslawa Porawska, Lukasz Porawski, Poznan
  - Katedra i Klinika Chorob Skornych i Wenerycznych, Pomorski Uniwersytet Medyczny, Szczecin
  - Spolka Cywilna Andrzej Krolicki, Tomasz Kochanowski "Laser Clinic", Szczecin
  - MTZ Clinical Research Sp. z o.o., Warsaw
  - Klinika Dermatologii, Warsaw
  - Zaklad Radiologii Lekarskiej, Warsaw
  - Katedra i Klinika Dermatologii, Wenerologii i Alergologii Akademii Medycznej we Wroclawiu, Wroclaw
  - Oddzial Dermatologiczny, Wroclaw
  - Poradnia Dermatologiczna, Wroclaw
- Grupo Dermatologico De Carolina (Office of Dr. Alma Cruz MD), Carolina, Puerto Rico
- Russia (10):
  - State Research Center of Dermatovenerology,, Moscow
  - State Research Center of Dermatovenerology, Moscow
  - Dermatovenerological dispensary #7, Moscow
  - Rostov-on-Don regional dermatovenerologic dispensary, Rostov-on-Don
  - Ryazan regional clinical dermatovenerologic dispensary, Ryazan
  - Dermatovenerologic dispensary #10 of Vyborg region, Saint Petersburg
  - Military Medical Academy N.A. S.M.Kirov, Saint Petersburg
  - North-Western State Medical University I.I. Mechnikov, Saint Petersburg
  - Smolensk State Medical Academy, Smolensk
  - Clinical hospital of emergency care N.V. Soloviev, Yaroslavl
- Serbia (2):
  - Clinical Hospital Center Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
- Singapore (2):
  - National Skin Centre, Singapore
  - Changi General Hospital, Singapore
- Slovakia (3):
  - Dermatovenerologicka klinika SZU, Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, Banská Bystrica
  - Oddelenie biologickej liecby, Narodny ustav reumatickych chorob, Piešťany
  - DOST-Dermatovenerologicke oddelenie sanatorneho typu, SANARE, spol. s r.o., Svidník
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Seoul
- Spain (6):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario La Princesa, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Sweden (6):
  - Hud kliniken- Skanes Universitetssjukhus i Malmo, Malmo, Sverige
  - Hudkliniken, Falun
  - Hermelinen Forskning AB, Luleå
  - Pharmacy: Sjukhusapoteket Lund, Lund
  - Hudkliniken, Stockholm
  - Karolinska University Hospital- Solna, Stockholm
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland
- Taiwan (6):
  - Chung Shan Medical University Hospital, Taichung, Taiwan Roc
  - Chang Gung Medical Foundation Kaohsiung Branch, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Taipei
  - Chang Gung Medical Foundation Linkou Branch, Taoyuan District
- Ukraine (8):
  - Dept of Dermatology and Venerology of SI "Crimean State Medical University n.a. S.I.Georgiyevskyy", Simferopol, Autonomous Republic of Crimea
  - Municipal Institution of health Care, Kharkiv
  - SI 'Institute for Dermatology and Venerology of AMS of Ukraine', Kharkiv
  - Kyiv Oleksandrivska Clin. Hosp., Dermatology department, NMU n.a. O.O. Bogomolets,, Kyiv
  - Dept of Dermatology and Venerology of Lugansk State Medical University,, Luhansk
  - Regional Municipal Dermatovenerologic Dispensary, Lviv
  - Dept of Dermatology and Venerology of ONMU, Odesa
  - Ternopil Regional Municipal Clinical Dermatovenerologic Dispensary, Ternopil
- United Kingdom (4):
  - Salford Royal NHS Foundation Trust, Salford, Manchester
  - Department of Dermatology, Nuneaton, Warwickshire
  - Whipps Cross University Hospital, London
  - eRT, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kristensen LE, Deodhar A, Leung YY, Vranic I, Mortezavi M, Fallon L, Yndestad A, Kinch CD, Gladman DD. Risk Stratification of Patients with Psoriatic Arthritis and Ankylosing Spondylitis for Treatment with Tofacitinib: A Review of Current Clinical Data. Rheumatol Ther. 2024 Jun;11(3):487-499. doi: 10.1007/s40744-024-00662-5. Epub 2024 May 2. PMID 38696034
- [Derived] Kristensen LE, Strober B, Poddubnyy D, Leung YY, Jo H, Kwok K, Vranic I, Fleishaker DL, Fallon L, Yndestad A, Gladman DD. Association between baseline cardiovascular risk and incidence rates of major adverse cardiovascular events and malignancies in patients with psoriatic arthritis and psoriasis receiving tofacitinib. Ther Adv Musculoskelet Dis. 2023 Feb 7;15:1759720X221149965. doi: 10.1177/1759720X221149965. eCollection 2023. PMID 36777695
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Valenzuela F, Korman NJ, Bissonnette R, Bakos N, Tsai TF, Harper MK, Ports WC, Tan H, Tallman A, Valdez H, Gardner AC. Tofacitinib in patients with moderate-to-severe chronic plaque psoriasis: long-term safety and efficacy in an open-label extension study. Br J Dermatol. 2018 Oct;179(4):853-862. doi: 10.1111/bjd.16798. Epub 2018 Aug 13. PMID 29782642
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921061&StudyName=A%20Long%20Term%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20Of%20CP-690%2C550%20For%20Patients%20With%20Moderate%20To%20Severe%20Chronic%20Plaque%20Psoriasi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2881 participants were enrolled in this study, however 2867 participants received treatment.
Groups:
- Tofacitinib 10 mg: Participants received Tofacitinib 10 milligram (mg) tablets orally twice daily from Day 1 until any safety finding requiring study discontinuation (up to a maximum of 66 months).
- Tofacitinib 5 mg or 10 mg: Participants received Tofacitinib 10 mg tablets orally twice daily for a period of 3 months. After 3 months of treatment, participants received twice daily dosing of tofacitinib 5 mg or 10 mg tablets until any safety and efficacy finding requiring study discontinuation (up to a maximum of 66 months). Dose adjustment (5 mg or 10 mg) was assessed on every 3 month visit and was based on investigator's discretion.
Period: Overall Study
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Started | 2281 | 586
Completed | 0 | 0
Not Completed | 2281 | 586
Not completed — Withdrawn Due to Pregnancy | 12 | 2
Not completed — Study Terminated by Sponsor | 978 | 349
Not completed — Protocol Violation | 43 | 12
Not completed — Withdrawal by Subject | 199 | 50
Not completed — Medication Error | 1 | 0
Not completed — Lost to Follow-up | 125 | 23
Not completed — Insufficient Clinical Response | 423 | 29
Not completed — Adverse Event | 300 | 78
Not completed — Death | 17 | 5
Not completed — Ongoing | 13 | 4
Not completed — Other Unspecified | 170 | 34

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg | Total
Number analyzed (Participants) | 2281 | 586 | 2867
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.5) | 47.0 (13.0) | 45.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 640 | 203 | 843
  Male | 1641 | 383 | 2024

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 4 weeks after last dose (up to 67 months) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2281 | 586
participants
  AEs | 1876 | 490
  SAEs | 304 | 88

2. Primary Outcome: Number of Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. AEs were classified according to the severity in 3 categories: a) mild: AEs did not interfere with participant's usual function; b) moderate: AEs interfered to some extent with participant's usual function; c) severe: AEs interfered significantly with participant's usual function.
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: adverse events
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2281 | 586
adverse events
  Mild | 5354 | 1749
  Moderate | 3268 | 766
  Severe | 410 | 136

3. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Abnormality criteria: hematology (hemoglobin, hematocrit, red blood cell <0.8*lower limit of normal [LLN]; reticulocyte<0.5*LLN,>1.5*ULN; platelets<0.5*LLN,>1.75* upper limit of normal [ULN]; WBC<0.6*LLN, >1.5*ULN; lymphocytes, neutrophils, basophils, eosinophils, monocytes<0.8*LLN; >1.2*ULN; coagulation (prothrombin [PT], PT ratio>1.1*ULN) liver function (bilirubin>1.5*ULN, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, gamma GT>0.3*ULN, protein, albumin<0.8*LLN; >1.2*ULN, globulin<0.5*LLN; >1.5*ULN); renal function (blood urea nitrogen, creatinine>1.3*ULN); electrolytes(sodium<0.95* LLN; >1.05* ULN, potassium, chloride, calcium, bicarbonate<0.9*LLN; >1.1*ULN), chemistry (glucose<0.6*LLN; >1.5* ULN), urinalysis (pH <4.5;>8, glucose, ketones, protein, blood, urobilinogen, nitrite, bilirubin, leukocyte esterase>=1; RBC, WBC>=20); lipids (cholesterol [C], LDL-C >1.3*ULN, HDL-C<0.8*LLN, triglycerides>1.3* ULN), hormones(T4, T3, T4, TSH<0.8* LLN; >1.2* ULN).
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2271 | 578
participants | 2203 | 565

4. Primary Outcome: Change From Baseline in Hemoglobin Level at Month 1
Time Frame: Baseline, Month 1
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'number of participants analyzed' signifies participants evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2277 | 586
gram per deciliter (g/dL)
  Baseline (n =2277, 586) | 14.64 (1.27) | 14.64 (1.24)
  Change at Month 1 (n =2201, 563) | -0.24 (0.83) | -0.32 (0.86)

5. Primary Outcome: Change From Baseline in Hemoglobin Level at Month 3
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2198 | 572
g/dL | -0.27 (0.85) | -0.39 (0.83)

6. Primary Outcome: Change From Baseline in Hemoglobin Level at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2051 | 563
g/dL | -0.27 (0.88) | -0.30 (0.87)

7. Primary Outcome: Change From Baseline in Hemoglobin Level at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1759 | 531
g/dL | -0.34 (0.93) | -0.30 (0.90)

8. Primary Outcome: Change From Baseline in Hemoglobin Level at Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1385 | 449
g/dL | -0.30 (0.96) | -0.29 (0.89)

9. Primary Outcome: Change From Baseline in Hemoglobin Level at Month 36
Time Frame: Baseline, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1114 | 380
g/dL | -0.32 (0.93) | -0.37 (0.88)

10. Primary Outcome: Change From Baseline in Hemoglobin Level at Month 48
Time Frame: Baseline, Month 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 415 | 127
g/dL | -0.35 (0.97) | -0.43 (0.94)

11. Primary Outcome: Change From Baseline in Lymphocyte and Neutrophil Count at Month 1
Time Frame: Baseline, Month 1
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2275 | 586
1000 cells/mm^3
  Baseline: Lymphocyte Count (n =2275, 586) | 1.76 (0.57) | 1.80 (0.56)
  Baseline: Neutrophil Count (n =2275, 586) | 4.74 (1.68) | 4.55 (1.70)
  Change at Month 1: Lymphocyte Count (n =2182, 559) | 0.07 (0.52) | 0.11 (0.56)
  Change at Month 1: Neutrophil Count (n =2182, 559) | -0.37 (1.65) | -0.48 (1.58)

12. Primary Outcome: Change From Baseline in Lymphocyte and Neutrophil Count at Month 3
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2183 | 570
1000 cells/mm^3
  Lymphocyte count | -0.00 (0.52) | 0.02 (0.52)
  Neutrophil Count | -0.28 (1.63) | -0.28 (1.60)

13. Primary Outcome: Change From Baseline in Lymphocyte and Neutrophil Count at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2034 | 559
1000 cells/mm^3
  Lymphocyte Count | -0.11 (0.51) | -0.05 (0.51)
  Neutrophil Count | -0.25 (1.61) | -0.22 (1.64)

14. Primary Outcome: Change From Baseline in Lymphocyte and Neutrophil Count at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1751 | 530
1000 cells/mm^3
  Lymphocyte Count | -0.21 (0.52) | -0.16 (0.48)
  Neutrophil Count | -0.23 (1.61) | -0.18 (1.58)

15. Primary Outcome: Change From Baseline in Lymphocyte and Neutrophil Count at Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1377 | 445
1000 cells/mm^3
  Lymphocyte Count | -0.28 (0.52) | -0.18 (0.54)
  Neutrophil Count | -0.19 (1.69) | -0.02 (1.59)

16. Primary Outcome: Change From Baseline in Lymphocyte and Neutrophil Count at Month 36
Time Frame: Baseline, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1111 | 377
1000 cells/mm^3
  Lymphocyte Count | -0.35 (0.55) | -0.24 (0.51)
  Neutrophil Count | -0.26 (1.61) | -0.11 (1.68)

17. Primary Outcome: Change From Baseline in Lymphocyte and Neutrophil Count at Month 48
Time Frame: Baseline, Month 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 413 | 127
1000 cells/mm^3
  Lymphocyte Count | -0.42 (0.52) | -0.27 (0.46)
  Neutrophil Count | -0.28 (1.70) | -0.07 (1.49)

18. Primary Outcome: Change From Baseline in Creatinine, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol (TC) Levels at Month 1
Time Frame: Baseline, Month 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2278 | 586
milligram per deciliter (mg/dL)
  Baseline: Creatinine (n =2278, 586) | 0.90 (0.17) | 0.88 (0.16)
  Baseline: LDL-C (n =2253, 585) | 114.14 (32.53) | 115.00 (35.03)
  Baseline: HDL-C (n =2277, 586) | 49.05 (13.93) | 51.87 (17.33)
  Baseline: TC (n =2277, 586) | 192.11 (38.10) | 194.96 (39.79)
  Change at Month 1: Creatinine (n =2204, 563) | 0.03 (0.10) | 0.02 (0.10)
  Change at Month 1: LDL-C (n =2125, 546) | 11.49 (28.77) | 11.55 (29.55)
  Change at Month 1: HDL-C (n =2203, 562) | 8.19 (9.89) | 8.63 (10.50)
  Change at Month 1: TC (n =2203, 562) | 21.12 (34.08) | 22.65 (34.36)

19. Primary Outcome: Change From Baseline in Creatinine, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol (TC) Levels at Month 3
Time Frame: Baseline, Month 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2211 | 573
mg/dL
  Creatinine (n =2211, 573) | 0.04 (0.21) | 0.03 (0.10)
  LDL-C (n =2130, 559) | 11.97 (29.77) | 10.44 (32.72)
  HDL-C (n =2204, 573) | 7.69 (10.23) | 7.96 (10.33)
  TC (n =2203, 573) | 21.52 (35.63) | 21.06 (38.34)

20. Primary Outcome: Change From Baseline in Creatinine, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol (TC) Levels at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2057 | 564
mg/dL
  Creatinine (n =2057, 564) | 0.03 (0.11) | 0.03 (0.10)
  LDL-C (n =1983, 553) | 11.44 (30.10) | 8.74 (33.22)
  HDL-C (n =2056, 564) | 7.68 (10.33) | 8.19 (11.60)
  TC (n =2057, 564) | 20.91 (35.94) | 19.17 (39.06)

21. Primary Outcome: Change From Baseline in Creatinine, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol (TC) Levels at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1777 | 533
mg/dL
  Creatinine (n =1777, 533) | 0.04 (0.12) | 0.04 (0.12)
  LDL-C (n =1728, 521) | 11.31 (31.45) | 9.65 (32.87)
  HDL-C (n =1776, 531) | 8.13 (10.48) | 6.88 (11.15)
  TC (n =1776, 531) | 21.20 (39.15) | 16.97 (37.84)

22. Primary Outcome: Change From Baseline in Creatinine, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol (TC) Levels at Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1398 | 450
mg/dL
  Creatinine (n =1398, 450) | 0.05 (0.11) | 0.04 (0.11)
  LDL-C (n =1353, 435) | 11.35 (35.33) | 10.13 (35.67)
  HDL-C (n =1397, 450) | 9.02 (11.62) | 7.55 (11.94)
  TC (n =1398, 450) | 21.74 (41.05) | 19.22 (39.69)

23. Primary Outcome: Change From Baseline in Creatinine, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol (TC) Levels at Month 36
Time Frame: Baseline, Month 36
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1122 | 384
mg/dL
  Creatinine (n =1122, 384) | 0.05 (0.12) | 0.04 (0.15)
  LDL-C (n =1085, 375) | 10.11 (35.83) | 7.25 (37.41)
  HDL-C (n =1119, 384) | 8.80 (11.59) | 6.39 (11.91)
  TC (n =1119, 384) | 20.20 (41.28) | 15.55 (43.59)

24. Primary Outcome: Change From Baseline in Creatinine, Low Density Lipoprotein Cholesterol (LDL-C), High Density Lipoprotein Cholesterol (HDL-C) and Total Cholesterol (TC) Levels at Month 48
Time Frame: Baseline, Month 48
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 417 | 127
mg/dL
  Creatinine (n =417, 127) | 0.04 (0.12) | 0.04 (0.11)
  LDL-C (n =402, 123) | 12.98 (36.89) | 6.61 (34.66)
  HDL-C (n =417, 127) | 8.62 (11.36) | 8.19 (12.72)
  TC (n =417, 127) | 24.99 (43.35) | 16.36 (40.99)

25. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) Levels at Month 1
Time Frame: Baseline, Month 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: international unit per liter (IU/L)
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2278 | 586
international unit per liter (IU/L)
  Baseline: AST (n =2278, 586) | 24.02 (12.22) | 24.66 (10.36)
  Baseline: ALT (n =2278, 586) | 28.47 (17.29) | 28.17 (16.56)
  Change at Month 1: AST (n =2198, 564) | 3.48 (15.39) | 4.07 (12.01)
  Change at Month 1: ALT (n =2199, 564) | 4.07 (19.04) | 4.84 (17.50)

26. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) Levels at Month 3
Time Frame: Baseline, Month 3
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2201 | 573
IU/L
  AST (n =2200, 573) | 4.09 (17.75) | 5.65 (16.37)
  ALT (n =2201, 573) | 4.86 (18.52) | 6.86 (20.80)

27. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) Levels at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2054 | 564
IU/L
  AST (n =2052, 564) | 4.50 (15.60) | 5.07 (14.90)
  ALT (n =2054, 564) | 5.98 (19.00) | 6.15 (18.40)

28. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) Levels at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1774 | 532
IU/L
  AST (n =1772, 531) | 4.88 (16.63) | 7.29 (22.70)
  ALT (n =1774, 532) | 6.68 (23.12) | 8.91 (25.21)

29. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) Levels at Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1398 | 450
IU/L
  AST (n =1397, 450) | 4.10 (14.64) | 6.77 (15.74)
  ALT (n =1398, 450) | 5.31 (19.37) | 7.56 (18.93)

30. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) Levels at Month 36
Time Frame: Baseline, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1122 | 384
IU/L
  AST | 5.38 (20.68) | 5.32 (15.65)
  ALT | 5.46 (20.61) | 6.56 (22.43)

31. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) Levels at Month 48
Time Frame: Baseline, Month 48
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 417 | 127
IU/L
  AST (n =416, 127) | 4.49 (14.05) | 8.40 (26.41)
  ALT (n =417, 127) | 4.92 (27.11) | 6.92 (20.98)

32. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Physical Examination
Description: Physical examinations included: general appearance; skin, head, eyes, ears, nose and throat; heart; lungs; abdomen; lower extremities (for the presence of peripheral edema) and lymph nodes. Clinical significance of change from baseline values in physical examination was based on investigator's discretion.
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2268 | 577
participants | 683 | 191

33. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Criteria for abnormalities in vital signs included: Systolic blood pressure (SBP): less than (<) 90 millimeter of mercury (mmHg) and maximum increase from baseline (IFB) of greater than or equal to (>=) 30 mmHg; diastolic blood pressure (DBP): <50 and greater than (>) 120 mmHg and maximum IFB of >=20 mmHg; heart rate: <40 and >120 beats per minute.
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2271 | 577
participants
  SBP (n =2271, 577) | 12 | 6
  DBP (n =2271, 577) | 12 | 1
  Heart Rate (n =2271, 577) | 3 | 1
  Maximum IFB in SBP (n =2267, 577) | 187 | 65
  Maximum IFB in DBP (n =2267, 577) | 221 | 74

34. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Month 1
Time Frame: Baseline, Month 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2277 | 586
millimeter of mercury (mmHg)
  Baseline: Systolic BP (n =2277, 586) | 126.07 (14.03) | 126.24 (14.12)
  Baseline: Diastolic BP (n =2277, 586) | 79.64 (9.42) | 78.88 (9.27)
  Change at Month 1: Systolic BP (n =2210, 564) | -0.43 (11.83) | -1.31 (11.55)
  Change at Month 1: Diastolic BP (n =2210, 564) | -0.03 (8.42) | 0.22 (8.45)

35. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Month 3
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2214 | 575
mmHg
  Systolic BP | -0.16 (11.97) | -0.95 (11.85)
  Diastolic BP | -0.26 (8.56) | 0.05 (8.52)

36. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2061 | 566
mmHg
  Systolic BP | 0.22 (12.18) | -0.15 (12.48)
  Diastolic BP | -0.05 (8.87) | 0.55 (8.74)

37. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1784 | 534
mmHg
  Systolic BP | 0.42 (11.97) | -0.20 (12.51)
  Diastolic BP | 0.23 (8.89) | 0.10 (9.10)

38. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1398 | 451
mmHg
  Systolic BP | 0.84 (13.00) | -0.07 (13.02)
  Diastolic BP | 0.36 (9.45) | 0.35 (8.85)

39. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Month 36
Time Frame: Baseline, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1123 | 386
mmHg
  Systolic BP | 0.52 (13.15) | 0.10 (13.92)
  Diastolic BP | 0.33 (9.33) | -0.06 (9.24)

40. Primary Outcome: Change From Baseline in Systolic Blood Pressure (BP) and Diastolic BP at Month 48
Time Frame: Baseline, Month 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 422 | 127
mmHg
  Systolic BP | 2.35 (13.45) | 1.13 (15.18)
  Diastolic BP | 0.97 (9.52) | 0.87 (9.80)

41. Primary Outcome: Change From Baseline in Heart Rate at Month 1
Time Frame: Baseline, Month 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2277 | 586
beats per minute
  Baseline (n =2277, 586) | 71.81 (9.67) | 71.46 (9.93)
  Change at Month 1 (n =2210, 563) | -0.82 (9.16) | -1.23 (9.03)

42. Primary Outcome: Change From Baseline in Heart Rate at Month 3
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2214 | 573
beats per minute | -0.57 (9.35) | -0.32 (9.19)

43. Primary Outcome: Change From Baseline in Heart Rate at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2061 | 565
beats per minute | -0.73 (9.65) | -1.05 (9.18)

44. Primary Outcome: Change From Baseline in Heart Rate at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1784 | 534
beats per minute | -1.13 (9.66) | -1.14 (9.07)

45. Primary Outcome: Change From Baseline in Heart Rate at Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1398 | 451
beats per minute | -1.07 (9.91) | -0.94 (8.89)

46. Primary Outcome: Change From Baseline in Heart Rate at Month 36
Time Frame: Baseline, Month 36
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1123 | 386
beats per minute | -1.38 (9.81) | -1.00 (9.26)

47. Primary Outcome: Change From Baseline in Heart Rate at Month 48
Time Frame: Baseline, Month 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 422 | 127
beats per minute | -0.91 (10.64) | -0.64 (10.64)

48. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Criteria for ECG abnormality: PR interval >=300 milliseconds (msec); QT interval >=500 msec; QTcB (Bazett's Correction) and QTcF (Fridericia's Correction) 450 to <480 msec, 480 to <500 msec and >=500 msec.
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2281 | 586
participants | 7 | 2

49. Primary Outcome: Change From Baseline in QRS Complex, PR, QT, QTcB, QTcF and RR Interval at Month 6
Time Frame: Baseline, Month 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2264 | 583
milliseconds (msec)
  Baseline: QRS Complex (n =2264, 583) | 92.88 (9.12) | 92.31 (9.75)
  Baseline: PR Interval (n =2258, 583) | 162.32 (21.32) | 158.91 (20.62)
  Baseline: QT Interval (n =2264, 583) | 392.39 (29.12) | 395.75 (29.70)
  Baseline: QTcB Interval (n =2264, 583) | 415.70 (23.83) | 416.91 (23.04)
  Baseline: QTcF Interval (n =2264, 583) | 407.48 (20.74) | 409.42 (20.11)
  Baseline: RR Interval (n =2264, 583) | 901.27 (145.58) | 911.59 (150.35)
  Change at Month 6: QRS Complex (n =1995, 550) | 1.51 (8.28) | 2.01 (7.50)
  Change at Month 6: PR Interval (n =1986, 549) | 2.46 (13.79) | 2.76 (14.81)
  Change at Month 6: QT Interval (n =1995, 550) | 2.25 (24.49) | 2.52 (24.39)
  Change at Month 6: QTcB Interval (n =1995, 550) | -0.84 (20.49) | -1.38 (20.31)
  Change at Month 6: QTcF Interval (n =1995, 550) | 0.23 (17.14) | -0.03 (17.68)
  Change at Month 6: RR Interval (n =1995, 550) | 14.35 (130.91) | 18.77 (123.49)

50. Primary Outcome: Change From Baseline in QRS Complex, PR, QT, QTcB, QTcF and RR Interval at Month 12
Time Frame: Baseline, Month 12
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1727 | 516
msec
  QRS Complex (n =1726, 516) | 1.89 (7.93) | 2.11 (7.53)
  PR Interval (n =1717, 515) | 2.80 (14.32) | 3.21 (14.31)
  QT Interval (n =1726, 516) | 2.49 (23.26) | 2.69 (23.00)
  QTcB Interval (n =1726, 516) | -1.04 (20.63) | -1.09 (20.83)
  QTcF Interval (n =1726, 516) | 0.16 (16.71) | 0.23 (17.20)
  RR Interval (n =1727, 516) | 15.94 (130.60) | 17.55 (128.16)

51. Primary Outcome: Change From Baseline in QRS Complex, PR, QT, QTcB, QTcF and RR Interval at Month 24
Time Frame: Baseline, Month 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 1352 | 432
msec
  QRS Complex (n =1352, 432) | 2.00 (8.55) | 2.42 (9.13)
  PR Interval (n =1346, 432) | 3.49 (14.55) | 3.81 (14.67)
  QT Interval (n =1352, 432) | 3.93 (24.93) | 2.28 (24.80)
  QTcB Interval (n =1352, 431) | 0.15 (20.77) | 0.78 (21.06)
  QTcF Interval (n =1352, 431) | 1.47 (16.86) | 1.25 (17.72)
  RR Interval (n =1352, 432) | 17.70 (139.47) | 8.66 (135.06)

52. Primary Outcome: Change From Baseline in QRS Complex, PR, QT, QTcB, QTcF and RR Interval at Month 36
Time Frame: Baseline, Month 36
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 845 | 283
msec
  QRS Complex (n =845, 283) | 1.75 (8.47) | 1.85 (10.37)
  PR Interval (n =840, 282) | 4.18 (14.50) | 3.25 (15.50)
  QT Interval (n =844, 283) | 4.31 (24.93) | 2.52 (22.63)
  QTcB Interval (n =844, 283) | 0.44 (21.29) | -0.01 (22.21)
  QTcF Interval (n =844, 283) | 1.79 (17.57) | 0.84 (17.63)
  RR Interval (n =845, 283) | 18.24 (136.44) | 15.14 (131.42)

53. Primary Outcome: Change From Baseline in QRS Complex, PR, QT, QTcB, QTcF and RR Interval at Month 48
Time Frame: Baseline, Month 48
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 126 | 55
msec
  QRS Complex (n =126, 55) | 2.37 (10.17) | 1.31 (5.37)
  PR Interval (n =126, 55) | 6.26 (12.58) | 1.98 (13.20)
  QT Interval (n =126, 55) | 6.43 (24.05) | 1.69 (23.43)
  QTcB Interval (n =125, 55) | 3.42 (20.11) | -2.00 (22.64)
  QTcF Interval (n =125, 55) | 4.55 (15.84) | -0.87 (19.38)
  RR Interval (n =126, 55) | 15.69 (143.06) | 20.78 (119.61)

54. Primary Outcome: Number of Participants With Adjudicated Cardiovascular Events
Description: Adjudicated cardiovascular events were assessed by adjudication committee as independent reviewers based on event documentation including: hospital discharge summaries, operative reports, clinic notes, ECGs, diagnostic enzymes, results of other diagnostic tests, autopsy reports and death certificate information; as applicable.
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2281 | 586
participants | 32 | 13

55. Primary Outcome: Number of Participants With Malignancy Events
Description: Malignancy events included lymphoma, and demyelinating neurologic events. Biopsies collected for malignancy events were submitted to the central laboratory for pathologist over-read.
Time Frame: Baseline up to 4 weeks after last dose of study drug (up to a maximum of 67 months)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2281 | 586
participants | 87 | 26

56. Secondary Outcome: Percentage of Participants Achieving Physician Global Assessment (PGA) Response of 'Clear' or 'Almost Clear'
Description: The PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema (E), induration (I), and scaling (S) across all psoriatic lesions in participants. The severity rating scores (Erythema: 0= no evidence of erythema to 4= dark, deep red; Induration: 0= no evidence of plaque elevation to 4= marked plaque elevation, hard/sharp borders; Scaling: 0= no evidence of scaling to 4= thick, coarse scale predominates) were summed (E + I + S = total) and the average (total/3) was taken. The total average was rounded to the nearest whole number score to determine the PGA. The 5-point scale for PGA was: 0= clear; 1= almost clear; 2= mild; 3= moderate; 4= severe, where higher score indicated more severity of psoriasis. Percentage of participants with response of 'clear' (score of '0') and 'almost clear' (score of '1') were reported.
Time Frame: Month 1, 3, 6, 12, 24, 36, 48
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study drug, excluding the participants who had compliance issues. Here, 'number of participants analyzed' signifies participants evaluable for this outcome measure and 'n' signifies participants who were evaluable at specified time points for each arm, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2200 | 571
percentage of participants
  Month 1 (n =2196, 563) | 50.36 [48.27 to 52.46] | 77.80 [74.36 to 81.23]
  Month 3 (n =2200, 571) | 54.86 [52.78 to 56.94] | 85.29 [82.38 to 88.19]
  Month 6 (n =2052, 564) | 54.97 [52.82 to 57.12] | 82.09 [78.93 to 85.26]
  Month 12 (n =1776, 532) | 54.79 [52.47 to 57.10] | 75.19 [71.52 to 78.86]
  Month 24 (n =1397, 448) | 54.62 [52.01 to 57.23] | 79.46 [75.72 to 83.20]
  Month 36 (n =1123, 385) | 57.35 [54.45 to 60.24] | 76.36 [72.12 to 80.61]
  Month 48 (n =422, 126) | 48.58 [43.81 to 53.35] | 77.78 [70.52 to 85.04]

57. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 75 Percent Reduction From Baseline in Psoriasis Area and Severity Index (PASI) Scores
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Each component of severity, that is, erythema, induration and scaling was assessed separately for four body areas (head and neck [h], upper limbs [u], trunk [t] and lower limbs [l]) on a 5-point scale ranging from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity. Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head and neck: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4. Percentage of participants with >=75 percent (%) reduction from baseline in PASI scores were reported.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: FAS included all participants who received at least 1 dose of study drug, excluding the participants who had compliance issues. Here, 'number of participants analyzed' signifies those participants who were evaluable for this outcome measure and 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2200 | 566
percentage of participants
  Month 1 (n =2194, 555) | 51.96 [49.87 to 54.05] | 71.89 [68.15 to 75.63]
  Month 3 (n =2200, 566) | 58.45 [56.40 to 60.51] | 84.45 [81.47 to 87.44]
  Month 6 (n =2048, 557) | 61.67 [59.56 to 63.78] | 86.00 [83.11 to 88.88]
  Month 12 (n =1775, 525) | 65.24 [63.02 to 67.45] | 80.76 [77.39 to 84.13]
  Month 24 (n =1393, 445) | 67.26 [64.80 to 69.73] | 84.94 [81.62 to 88.27]
  Month 36 (n =1118, 380) | 70.75 [68.08 to 73.42] | 83.95 [80.26 to 87.64]
  Month 48 (n =422, 124) | 64.93 [60.38 to 69.48] | 83.06 [76.46 to 89.67]

58. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Scores
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Each component of severity, that is, erythema, induration and scaling was assessed separately for four body areas (head and neck [h], upper limbs [u], trunk [t] and lower limbs [l]) on a 5-point scale ranging from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity. Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head and neck: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2266 | 585
units on a scale
  Baseline (n =2266, 585) | 21.85 (9.48) | 19.05 (8.89)
  Month 1 (n =2198, 561) | 6.60 (7.14) | 3.09 (4.81)
  Month 3 (n =2205, 572) | 5.64 (6.33) | 1.95 (3.25)
  Month 6 (n =2051, 563) | 5.31 (6.31) | 1.90 (3.25)
  Month 12 (n =1779, 531) | 4.72 (5.29) | 2.38 (3.57)
  Month 24 (n =1397, 449) | 4.41 (5.08) | 1.90 (2.65)
  Month 36 (n =1121, 384) | 3.91 (4.66) | 2.19 (3.23)
  Month 48 (n =422, 126) | 4.75 (5.37) | 1.85 (2.31)

59. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Scores at Month 1, 3, 6, 12, 24, 36 and 48
Description: as for outcome 58
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2201 | 572
units on a scale
  Month 1 (n =2195, 561) | -15.26 (9.96) | -16.00 (9.57)
  Month 3 (n =2201, 572) | -16.18 (9.73) | -16.99 (9.27)
  Month 6 (n =2049, 563) | -16.56 (9.54) | -17.03 (9.16)
  Month 12 (n =1776, 531) | -17.01 (9.33) | -16.45 (9.04)
  Month 24 (n =1394, 449) | -17.25 (9.35) | -16.67 (8.70)
  Month 36 (n =1119, 384) | -17.44 (9.23) | -16.49 (8.81)
  Month 48 (n =422, 126) | -16.16 (8.61) | -15.47 (9.04)

60. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Component Scores: Erythema
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Erythema was assessed separately for four body areas (head and neck, upper limbs, trunk and lower limbs) on a 5-point scale ranges from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2266 | 585
units on a scale
  Baseline: Head/Neck (n =2266, 585) | 2.26 (0.99) | 2.13 (1.08)
  Month 1: Head/Neck (n =2198, 561) | 0.82 (0.96) | 0.47 (0.81)
  Month 3: Head/Neck (n =2205, 572) | 0.76 (0.95) | 0.34 (0.65)
  Month 6: Head/Neck (n =2051, 563) | 0.75 (0.95) | 0.42 (0.75)
  Month 12: Head/Neck (n =1779, 531) | 0.70 (0.92) | 0.49 (0.82)
  Month 24: Head/Neck (n =1397, 449) | 0.66 (0.93) | 0.47 (0.75)
  Month 36: Head/Neck (n =1121, 384) | 0.57 (0.88) | 0.48 (0.79)
  Month 48: Head/Neck (n =422, 126) | 0.70 (0.93) | 0.34 (0.69)
  Baseline: Upper Limbs (n =2266, 585) | 2.82 (0.74) | 2.68 (0.86)
  Month 1: Upper Limbs (n =2198, 561) | 1.29 (0.98) | 0.71 (0.86)
  Month 3: Upper Limbs (n =2205, 572) | 1.23 (1.00) | 0.57 (0.79)
  Month 6: Upper Limbs (n =2051, 563) | 1.20 (1.01) | 0.58 (0.83)
  Month 12: Upper Limbs (n =1779, 531) | 1.16 (1.01) | 0.74 (0.95)
  Month 24: Upper Limbs (n =1397, 449) | 1.13 (1.03) | 0.61 (0.85)
  Month 36: Upper Limbs (n =1121, 384) | 1.06 (1.01) | 0.68 (0.86)
  Month 48: Upper Limbs (n =422, 126) | 1.18 (1.03) | 0.58 (0.84)
  Baseline: Trunk (n =2266, 585) | 2.83 (0.83) | 2.73 (0.94)
  Month 1: Trunk (n =2198, 561) | 1.18 (1.11) | 0.62 (0.92)
  Month 3: Trunk (n =2205, 572) | 1.06 (1.09) | 0.41 (0.73)
  Month 6: Trunk (n =2051, 563) | 1.03 (1.09) | 0.41 (0.79)
  Month 12: Trunk (n =1779, 531) | 0.99 (1.08) | 0.51 (0.89)
  Month 24: Trunk (n =1397, 449) | 0.96 (1.08) | 0.49 (0.84)
  Month 36: Trunk (n =1121, 384) | 0.86 (1.06) | 0.53 (0.90)
  Month 48: Trunk (n =422, 126) | 1.00 (1.10) | 0.50 (0.86)
  Baseline: Lower Limbs (n =2266, 585) | 3.10 (0.70) | 2.94 (0.89)
  Month 1: Lower Limbs (n =2198, 561) | 1.37 (1.09) | 0.79 (0.95)
  Month 3: Lower Limbs (n =2205, 572) | 1.24 (1.08) | 0.58 (0.84)
  Month 6: Lower Limbs (n =2051, 563) | 1.20 (1.11) | 0.52 (0.81)
  Month 12: Lower Limbs (n =1779, 531) | 1.17 (1.10) | 0.69 (0.98)
  Month 24: Lower Limbs (n =1397, 449) | 1.15 (1.11) | 0.59 (0.90)
  Month 36: Lower Limbs (n =1121, 384) | 1.07 (1.11) | 0.67 (0.96)
  Month 48: Lower Limbs (n =422, 126) | 1.20 (1.11) | 0.61 (0.91)

61. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Component Scores: Induration
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Induration was assessed separately for four body areas (head and neck, upper limbs, trunk and lower limbs) on a 5-point scale ranges from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2266 | 585
units on a scale
  Baseline: Head/Neck (n =2266, 585) | 1.97 (1.01) | 1.88 (1.10)
  Month 1: Head/Neck (n =2198, 561) | 0.65 (0.85) | 0.35 (0.73)
  Month 3: Head/Neck (n =2205, 572) | 0.60 (0.84) | 0.26 (0.56)
  Month 6: Head/Neck (n =2051, 563) | 0.59 (0.86) | 0.31 (0.67)
  Month 12: Head/Neck (n =1779, 531) | 0.55 (0.81) | 0.38 (0.71)
  Month 24: Head/Neck (n =1397, 449) | 0.53 (0.82) | 0.37 (0.68)
  Month 36: Head/Neck (n =1121, 384) | 0.46 (0.77) | 0.37 (0.68)
  Month 48: Head/Neck (n =422, 126) | 0.60 (0.85) | 0.26 (0.60)
  Baseline: Upper Limbs (n =2266, 585) | 2.64 (0.77) | 2.50 (0.93)
  Month 1: Upper Limbs (n =2198, 561) | 1.21 (0.99) | 0.66 (0.88)
  Month 3: Upper Limbs (n =2205, 572) | 1.17 (1.01) | 0.53 (0.81)
  Month 6: Upper Limbs (n =2051, 563) | 1.15 (1.02) | 0.55 (0.85)
  Month 12: Upper Limbs (n =1779, 531) | 1.11 (1.01) | 0.69 (0.95)
  Month 24: Upper Limbs (n =1397, 449) | 1.08 (1.02) | 0.53 (0.84)
  Month 36: Upper Limbs (n =1121, 384) | 1.00 (1.01) | 0.60 (0.82)
  Month 48: Upper Limbs (n =422, 126) | 1.09 (1.00) | 0.50 (0.75)
  Baseline: Trunk (n =2266, 585) | 2.57 (0.86) | 2.51 (1.01)
  Month 1: Trunk (n =2198, 561) | 1.02 (1.04) | 0.52 (0.86)
  Month 3: Trunk (n =2205, 572) | 0.91 (1.02) | 0.34 (0.68)
  Month 6: Trunk (n =2051, 563) | 0.88 (1.00) | 0.34 (0.71)
  Month 12: Trunk (n =1779, 531) | 0.87 (1.00) | 0.42 (0.77)
  Month 24: Trunk (n =1397, 449) | 0.82 (0.98) | 0.39 (0.73)
  Month 36: Trunk (n =1121, 384) | 0.75 (0.97) | 0.43 (0.79)
  Month 48: Trunk (n =422, 126) | 0.91 (1.05) | 0.44 (0.80)
  Baseline: Lower Limbs (n =2266, 585) | 2.85 (0.76) | 2.77 (0.96)
  Month 1: Lower Limbs (n =2198, 561) | 1.22 (1.04) | 0.68 (0.95)
  Month 3: Lower Limbs (n =2205, 572) | 1.10 (1.04) | 0.51 (0.84)
  Month 6: Lower Limbs (n =2051, 563) | 1.08 (1.06) | 0.47 (0.82)
  Month 12: Lower Limbs (n =1779, 531) | 1.05 (1.03) | 0.61 (0.94)
  Month 24: Lower Limbs (n =1397, 449) | 1.02 (1.03) | 0.49 (0.83)
  Month 36: Lower Limbs (n =1121, 384) | 0.95 (1.03) | 0.57 (0.87)
  Month 48: Lower Limbs (n =422, 126) | 1.07 (1.04) | 0.48 (0.79)

62. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Component Scores: Scaling
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Scaling was assessed separately for four body areas (head and neck, upper limbs, trunk and lower limbs) on a 5-point scale ranges from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2266 | 585
units on a scale
  Baseline: Head/Neck (n =2266, 585) | 2.22 (1.08) | 2.10 (1.11)
  Month 1: Head/Neck (n =2198, 561) | 0.75 (0.95) | 0.42 (0.79)
  Month 3: Head/Neck (n =2205, 572) | 0.71 (0.95) | 0.32 (0.66)
  Month 6: Head/Neck (n =2051, 563) | 0.71 (0.97) | 0.40 (0.77)
  Month 12: Head/Neck (n =1779, 531) | 0.67 (0.92) | 0.48 (0.84)
  Month 24: Head/Neck (n =1397, 449) | 0.60 (0.88) | 0.45 (0.77)
  Month 36: Head/Neck (n =1121, 384) | 0.55 (0.88) | 0.47 (0.79)
  Month 48: Head/Neck (n =422, 126) | 0.65 (0.93) | 0.34 (0.72)
  Baseline: Upper Limbs (n =2266, 585) | 2.65 (0.82) | 2.52 (0.96)
  Month 1: Upper Limbs (n =2198, 561) | 1.22 (1.01) | 0.69 (0.89)
  Month 3: Upper Limbs (n =2205, 572) | 1.18 (1.04) | 0.55 (0.80)
  Month 6: Upper Limbs (n =2051, 563) | 1.16 (1.05) | 0.58 (0.87)
  Month 12: Upper Limbs (n =1779, 531) | 1.12 (1.03) | 0.72 (0.97)
  Month 24: Upper Limbs (n =1397, 449) | 1.08 (1.03) | 0.58 (0.84)
  Month 36: Upper Limbs (n =1121, 384) | 1.01 (1.02) | 0.62 (0.83)
  Month 48: Upper Limbs (n =422, 126) | 1.13 (1.09) | 0.53 (0.79)
  Baseline: Trunk (n =2266, 585) | 2.55 (0.89) | 2.47 (1.00)
  Month 1: Trunk (n =2198, 561) | 0.97 (1.02) | 0.50 (0.83)
  Month 3: Trunk (n =2205, 572) | 0.87 (1.00) | 0.33 (0.64)
  Month 6: Trunk (n =2051, 563) | 0.85 (0.99) | 0.33 (0.70)
  Month 12: Trunk (n =1779, 531) | 0.83 (0.97) | 0.40 (0.76)
  Month 24: Trunk (n =1397, 449) | 0.78 (0.95) | 0.39 (0.72)
  Month 36: Trunk (n =1121, 384) | 0.71 (0.93) | 0.42 (0.77)
  Month 48: Trunk (n =422, 126) | 0.86 (0.99) | 0.40 (0.78)
  Baseline: Lower Limbs (n =2266, 585) | 2.89 (0.81) | 2.79 (1.00)
  Month 1: Lower Limbs (n =2198, 561) | 1.23 (1.08) | 0.70 (0.93)
  Month 3: Lower Limbs (n =2205, 572) | 1.12 (1.08) | 0.48 (0.78)
  Month 6: Lower Limbs (n =2051, 563) | 1.11 (1.10) | 0.48 (0.83)
  Month 12: Lower Limbs (n =1779, 531) | 1.07 (1.07) | 0.64 (0.98)
  Month 24: Lower Limbs (n =1397, 449) | 1.04 (1.06) | 0.53 (0.84)
  Month 36: Lower Limbs (n =1121, 384) | 0.94 (1.03) | 0.60 (0.90)
  Month 48: Lower Limbs (n =422, 126) | 1.09 (1.09) | 0.48 (0.76)

63. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Component Scores: Erythema at Month 1, 3, 6, 12, 24, 36 and 48
Description: as for outcome 60
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2201 | 572
units on a scale
  Month 1: Head/Neck (n =2195, 561) | -1.43 (1.15) | -1.66 (1.20)
  Month 3: Head/Neck (n =2201, 572) | -1.50 (1.18) | -1.80 (1.18)
  Month 6: Head/Neck (n =2049, 563) | -1.52 (1.20) | -1.72 (1.21)
  Month 12: Head/Neck (n =1776, 531) | -1.56 (1.19) | -1.64 (1.22)
  Month 24: Head/Neck (n =1394, 449) | -1.62 (1.19) | -1.67 (1.23)
  Month 36: Head/Neck (n =1119, 384) | -1.72 (1.18) | -1.67 (1.20)
  Month 48: Head/Neck (n =422, 126) | -1.55 (1.19) | -1.70 (1.13)
  Month 1: Upper Limbs (n =2195, 561) | -1.53 (1.12) | -1.98 (1.18)
  Month 3: Upper Limbs (n =2201, 572) | -1.59 (1.15) | -2.12 (1.14)
  Month 6: Upper Limbs (n =2049, 563) | -1.62 (1.15) | -2.09 (1.13)
  Month 12: Upper Limbs (n =1776, 531) | -1.67 (1.15) | -1.94 (1.21)
  Month 24: Upper Limbs (n =1394, 449) | -1.70 (1.18) | -2.05 (1.19)
  Month 36: Upper Limbs (n =1119, 384) | -1.78 (1.17) | -2.00 (1.18)
  Month 48: Upper Limbs (n =422, 126) | -1.62 (1.16) | -1.90 (1.22)
  Month 1: Trunk (n =2195, 561) | -1.65 (1.22) | -2.12 (1.26)
  Month 3: Trunk (n =2201, 572) | -1.77 (1.24) | -2.33 (1.17)
  Month 6: Trunk (n =2049, 563) | -1.81 (1.24) | -2.32 (1.19)
  Month 12: Trunk (n =1776, 531) | -1.86 (1.24) | -2.21 (1.25)
  Month 24: Trunk (n =1394, 449) | -1.88 (1.25) | -2.22 (1.26)
  Month 36: Trunk (n =1119, 384) | -1.99 (1.26) | -2.18 (1.30)
  Month 48: Trunk (n =422, 126) | -1.82 (1.22) | -2.08 (1.17)
  Month 1: Lower Limbs (n =2195, 561) | -1.72 (1.19) | -2.16 (1.26)
  Month 3: Lower Limbs (n =2201, 572) | -1.87 (1.21) | -2.36 (1.21)
  Month 6: Lower Limbs (n =2049, 563) | -1.90 (1.22) | -2.42 (1.18)
  Month 12: Lower Limbs (n =1776, 531) | -1.94 (1.23) | -2.24 (1.33)
  Month 24: Lower Limbs (n =1394, 449) | -1.95 (1.25) | -2.32 (1.24)
  Month 36: Lower Limbs (n =1119, 384) | -2.04 (1.23) | -2.28 (1.30)
  Month 48: Lower Limbs (n =422, 126) | -1.87 (1.20) | -2.17 (1.21)

64. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Component Scores: Induration at Month 1, 3, 6, 12, 24, 36 and 48
Description: as for outcome 61
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2201 | 572
units on a scale
  Month 1: Head/Neck (n =2195, 561) | -1.32 (1.13) | -1.53 (1.15)
  Month 3: Head/Neck (n =2201, 572) | -1.37 (1.17) | -1.63 (1.14)
  Month 6: Head/Neck (n =2049, 563) | -1.40 (1.16) | -1.57 (1.18)
  Month 12: Head/Neck (n =1776, 531) | -1.44 (1.18) | -1.49 (1.18)
  Month 24: Head/Neck (n =1394, 449) | -1.48 (1.17) | -1.51 (1.21)
  Month 36: Head/Neck (n =1119, 384) | -1.55 (1.17) | -1.51 (1.15)
  Month 48: Head/Neck (n =422, 126) | -1.35 (1.17) | -1.41 (1.10)
  Month 1: Upper Limbs (n =2195, 561) | -1.43 (1.14) | -1.85 (1.22)
  Month 3: Upper Limbs (n =2201, 572) | -1.47 (1.17) | -1.97 (1.16)
  Month 6: Upper Limbs (n =2049, 563) | -1.49 (1.15) | -1.94 (1.19)
  Month 12: Upper Limbs (n =1776, 531) | -1.54 (1.14) | -1.82 (1.27)
  Month 24: Upper Limbs (n =1394, 449) | -1.57 (1.18) | -1.97 (1.19)
  Month 36: Upper Limbs (n =1119, 384) | -1.65 (1.17) | -1.92 (1.18)
  Month 48: Upper Limbs (n =422, 126) | -1.53 (1.14) | -1.83 (1.14)
  Month 1: Trunk (n =2195, 561) | -1.55 (1.19) | -2.01 (1.26)
  Month 3: Trunk (n =2201, 572) | -1.65 (1.22) | -2.17 (1.18)
  Month 6: Trunk (n =2049, 563) | -1.70 (1.19) | -2.18 (1.20)
  Month 12: Trunk (n =1776, 531) | -1.71 (1.20) | -2.10 (1.24)
  Month 24: Trunk (n =1394, 449) | -1.76 (1.19) | -2.13 (1.20)
  Month 36: Trunk (n =1119, 384) | -1.85 (1.20) | -2.09 (1.23)
  Month 48: Trunk (n =422, 126) | -1.68 (1.17) | -1.87 (1.20)
  Month 1: Lower Limbs (n =2195, 561) | -1.63 (1.22) | -2.09 (1.31)
  Month 3: Lower Limbs (n =2201, 572) | -1.75 (1.22) | -2.26 (1.24)
  Month 6: Lower Limbs (n =2049, 563) | -1.78 (1.23) | -2.30 (1.23)
  Month 12: Lower Limbs (n =1776, 531) | -1.82 (1.20) | -2.17 (1.33)
  Month 24: Lower Limbs (n =1394, 449) | -1.85 (1.22) | -2.28 (1.24)
  Month 36: Lower Limbs (n =1119, 384) | -1.93 (1.21) | -2.22 (1.29)
  Month 48: Lower Limbs (n =422, 126) | -1.77 (1.18) | -2.07 (1.24)

65. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Component Scores: Scaling at Month 1, 3, 6, 12, 24, 36 and 48
Description: as for outcome 62
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2201 | 572
units on a scale
  Month 1: Head/Neck (n =2195, 561) | -1.46 (1.19) | -1.69 (1.20)
  Month 3: Head/Neck (n =2201, 572) | -1.51 (1.24) | -1.78 (1.19)
  Month 6: Head/Neck (n =2049, 563) | -1.52 (1.24) | -1.70 (1.22)
  Month 12: Head/Neck (n =1776, 531) | -1.56 (1.25) | -1.61 (1.24)
  Month 24: Head/Neck (n =1394, 449) | -1.63 (1.24) | -1.63 (1.27)
  Month 36: Head/Neck (n =1119, 384) | -1.68 (1.22) | -1.64 (1.22)
  Month 48: Head/Neck (n =422, 126) | -1.53 (1.24) | -1.58 (1.17)
  Month 1: Upper Limbs (n =2195, 561) | -1.44 (1.18) | -1.84 (1.24)
  Month 3: Upper Limbs (n =2201, 572) | -1.47 (1.20) | -1.97 (1.18)
  Month 6: Upper Limbs (n =2049, 563) | -1.49 (1.21) | -1.94 (1.26)
  Month 12: Upper Limbs (n =1776, 531) | -1.52 (1.21) | -1.82 (1.30)
  Month 24: Upper Limbs (n =1394, 449) | -1.56 (1.22) | -1.96 (1.22)
  Month 36: Upper Limbs (n =1119, 384) | -1.65 (1.19) | -1.93 (1.15)
  Month 48: Upper Limbs (n =422, 126) | -1.45 (1.19) | -1.78 (1.22)
  Month 1: Trunk (n =2195, 561) | -1.58 (1.20) | -1.98 (1.24)
  Month 3: Trunk (n =2201, 572) | -1.67 (1.22) | -2.14 (1.14)
  Month 6: Trunk (n =2049, 563) | -1.70 (1.19) | -2.14 (1.22)
  Month 12: Trunk (n =1776, 531) | -1.72 (1.21) | -2.08 (1.23)
  Month 24: Trunk (n =1394, 449) | -1.77 (1.20) | -2.11 (1.19)
  Month 36: Trunk (n =1119, 384) | -1.84 (1.20) | -2.06 (1.23)
  Month 48: Trunk (n =422, 126) | -1.62 (1.19) | -1.80 (1.18)
  Month 1: Lower Limbs (n =2195, 561) | -1.67 (1.24) | -2.09 (1.30)
  Month 3: Lower Limbs (n =2201, 572) | -1.77 (1.26) | -2.30 (1.23)
  Month 6: Lower Limbs (n =2049, 563) | -1.79 (1.27) | -2.30 (1.25)
  Month 12: Lower Limbs (n =1776, 531) | -1.83 (1.26) | -2.15 (1.36)
  Month 24: Lower Limbs (n =1394, 449) | -1.86 (1.27) | -2.25 (1.24)
  Month 36: Lower Limbs (n =1119, 384) | -1.97 (1.23) | -2.21 (1.26)
  Month 48: Lower Limbs (n =422, 126) | -1.77 (1.29) | -2.11 (1.23)

66. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 50 Percent Reduction From Baseline in Psoriasis Area and Severity Index (PASI) Scores
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Each component of severity, that is, erythema, induration and scaling was assessed separately for four body areas (head and neck [h], upper limbs [u], trunk [t] and lower limbs [l]) on a 5-point scale ranging from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity. Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head and neck: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4. Percentage of participants with >=50% reduction from baseline in PASI scores were reported.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2200 | 566
percentage of participants
  Month 1 (n =2194, 555) | 76.53 [74.75 to 78.30] | 86.67 [83.84 to 89.49]
  Month 3 (n =2200, 566) | 81.59 [79.97 to 83.21] | 95.05 [93.27 to 96.84]
  Month 6 (n =2048, 557) | 85.64 [84.13 to 87.16] | 93.90 [91.91 to 95.88]
  Month 12 (n =1775, 525) | 87.66 [86.13 to 89.19] | 93.14 [90.98 to 95.30]
  Month 24 (n =1393, 445) | 88.87 [87.22 to 90.52] | 94.61 [92.51 to 96.71]
  Month 36 (n =1118, 380) | 90.97 [89.29 to 92.65] | 92.63 [90.00 to 95.26]
  Month 48 (n =422, 124) | 88.86 [85.86 to 91.86] | 97.58 [94.88 to 100.00]

67. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 90 Percent Reduction From Baseline in Psoriasis Area and Severity Index (PASI) Scores
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Each component of severity, that is, erythema, induration and scaling was assessed separately for four body areas (head and neck [h], upper limbs [u], trunk [t] and lower limbs [l]) on a 5-point scale ranging from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity. Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head and neck: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4. Percentage of participants with >=90% reduction from baseline in PASI scores were reported.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2200 | 566
percentage of participants
  Month 1 (n =2194, 555) | 29.99 [28.07 to 31.91] | 56.04 [51.91 to 60.17]
  Month 3 (n =2200, 566) | 33.73 [31.75 to 35.70] | 65.37 [61.45 to 69.29]
  Month 6 (n =2048, 557) | 35.21 [33.14 to 37.27] | 65.89 [61.95 to 69.83]
  Month 12 (n =1775, 525) | 35.94 [33.71 to 38.18] | 61.71 [57.56 to 65.87]
  Month 24 (n =1393, 445) | 38.33 [35.78 to 40.89] | 62.02 [57.51 to 66.53]
  Month 36 (n =1118, 380) | 43.02 [40.12 to 45.93] | 60.53 [55.61 to 65.44]
  Month 48 (n =422, 124) | 34.36 [29.83 to 38.89] | 58.06 [49.38 to 66.75]

68. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 125 Percent Increase From Baseline in Psoriasis Area and Severity Index (PASI) Scores
Description: PASI score is the combined assessment of lesion severity (estimated by 3 components: of erythema, induration and scaling) and area affected into single score range: 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. Each component of severity, that is, erythema, induration and scaling was assessed separately for four body areas (head and neck [h], upper limbs [u], trunk [t] and lower limbs [l]) on a 5-point scale ranging from 0=no involvement, 1=slight, 2=moderate, 3=marked, 4=very marked. Higher score indicates greater severity. Final PASI score = 0.1Ah (Eh + Ih + Sh) + 0.2Au (Eu + Iu + Su) + 0.3At (Et + It + St) + 0.4Al (El + Il + Sl), where head and neck: 0.1; upper limbs: 0.2; trunk: 0.3; lower limbs: 0.4. Percentage of participants with >=125% increase from baseline in PASI scores were reported.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2200 | 566
percentage of participants
  Month 1 (n =2194, 555) | 0.96 [0.55 to 1.36] | 1.08 [0.22 to 1.94]
  Month 3 (n =2200, 566) | 1.18 [0.73 to 1.63] | 0.71 [0.02 to 1.40]
  Month 6 (n =2048, 557) | 1.27 [0.78 to 1.75] | 0.90 [0.11 to 1.68]
  Month 12 (n =1775, 525) | 0.90 [0.46 to 1.34] | 1.33 [0.35 to 2.31]
  Month 24 (n =1393, 445) | 0.93 [0.43 to 1.44] | 0.90 [0.02 to 1.78]
  Month 36 (n =1118, 380) | 0.54 [0.11 to 0.96] | 1.32 [0.17 to 2.46]
  Month 48 (n =422, 124) | 0.71 [0.00 to 1.51] | 0.00 [0.00 to 0.00]

69. Secondary Outcome: Itch Severity Item (ISI) Scores
Description: ISI assessed severity of itching due to psoriasis. ISI was a single item, horizontal numeric rating scale. Participants were asked to rate their 'severity of itching' due to psoriasis over the past 24 hours on a numeric rating scale anchored by the terms '0=no itching' and '10=worst possible itching' at the ends. Higher scores indicated greater severity of itching.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2197 | 572
units on a scale
  Baseline (n =2172, 566) | 5.76 (2.91) | 5.17 (3.00)
  Month 1 (n =2196, 561) | 1.88 (2.26) | 0.92 (1.53)
  Month 3 (n =2197, 572) | 1.83 (2.32) | 0.72 (1.39)
  Month 6 (n =2047, 560) | 1.87 (2.33) | 0.82 (1.51)
  Month 12 (n =1774, 530) | 1.79 (2.21) | 1.08 (1.67)
  Month 24 (n =1394, 449) | 1.83 (2.23) | 1.01 (1.54)
  Month 36 (n =1117, 383) | 1.69 (2.12) | 1.21 (1.72)
  Month 48 (n =417, 127) | 1.92 (2.30) | 1.24 (1.74)

70. Secondary Outcome: Change From Baseline in Itch Severity Item (ISI) Scores at Month 1, 3, 6, 12, 24, 36 and 48
Description: as for outcome 69
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2107 | 554
units on a scale
  Month 1 (n =2107, 544) | -3.88 (3.06) | -4.26 (3.07)
  Month 3 (n =2103, 554) | -3.94 (3.18) | -4.44 (3.06)
  Month 6 (n =1958, 543) | -3.91 (3.20) | -4.36 (3.14)
  Month 12 (n =1693, 514) | -3.90 (3.17) | -4.01 (3.30)
  Month 24 (n =1340, 435) | -3.80 (3.14) | -4.11 (3.17)
  Month 36 (n =1078, 372) | -3.95 (3.18) | -3.84 (3.06)
  Month 48 (n =411, 126) | -4.03 (3.19) | -3.78 (3.25)

71. Secondary Outcome: Dermatology Life Quality Index (DLQI) Scores
Description: The DLQI was a validated, self-administered, 10-item quality-of-life questionnaire that consisted of 10 items that assessed the impact of skin disease on quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). Each question was scored on a scale of 0=not at all/not relevant to 3=very much. Response from all of the 10 questions were added to derive the DLQI total scores. Total DLQI scores ranges from 0=not at all to 30=very much, with higher scores indicating greater impairment in quality of life.
Time Frame: Baseline, Month 1, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2243 | 582
units on a scale
  Baseline (n =2243, 582) | 12.73 (7.12) | 10.95 (6.61)
  Month 1 (n =2189, 559) | 4.11 (5.23) | 2.14 (3.43)
  Month 6 (n =2028, 557) | 3.68 (5.00) | 1.67 (3.33)
  Month 12 (n =1751, 528) | 3.44 (4.65) | 1.71 (2.92)
  Month 24 (n =1361, 441) | 3.49 (4.71) | 1.94 (3.29)
  Month 36 (n =1093, 372) | 2.97 (4.05) | 1.98 (3.35)
  Month 48 (n =407, 124) | 3.20 (4.39) | 1.81 (2.98)

72. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Scores at Month 1, 6, 12, 24, 36 and 48
Description: as for outcome 71
Time Frame: Baseline, Month 1, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2163 | 556
units on a scale
  Month 1 (n =2163, 556) | -8.61 (7.00) | -8.75 (6.56)
  Month 6 (n =2005, 554) | -9.14 (7.06) | -9.22 (6.92)
  Month 12 (n =1730, 525) | -9.23 (6.91) | -9.02 (6.68)
  Month 24 (n =1345, 438) | -9.08 (6.82) | -8.47 (6.43)
  Month 36 (n =1083, 369) | -9.47 (6.80) | -8.46 (6.14)
  Month 48 (n =404, 122) | -8.99 (6.74) | -7.78 (6.10)

73. Secondary Outcome: 36-Item Short-Form (SF-36) Health Survey Version 2, Acute: Physical Component Summary Scores
Description: The SF-36 questionnaire, version 2, acute was a 36-item generic health status measure. SF-36 evaluated 8 health-related aspects of an individual: physical functioning, role-physical, bodily pain, social functioning, mental health, role emotional, vitality, and general health. The score range for each of the 8 health aspects ranged from 0 (worst) to 100 (best), with higher scores indicating good health condition. Two summary scale scores were computed from the 8 health aspect scores: physical component summary score and mental component summary score. Score range for both summary scales ranged from 0 (worst) to 100 (best), with higher scores indicating good health condition.
Time Frame: Baseline, Month 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2233 | 580
units on a scale
  Baseline (n =2233, 580) | 47.31 (9.38) | 48.94 (9.12)
  Month 6 (n =2025, 557) | 51.78 (8.24) | 53.51 (7.30)
  Month 12 (n =1750, 524) | 51.96 (8.13) | 53.58 (7.19)
  Month 24 (n =1362, 442) | 51.91 (7.80) | 53.15 (7.32)
  Month 36 (n =857, 286) | 52.01 (8.08) | 53.05 (7.28)
  Month 48 (n =124, 56) | 52.93 (6.79) | 52.36 (8.39)

74. Secondary Outcome: 36-Item Short-Form (SF-36) Health Survey Version 2, Acute: Mental Component Summary Scores
Description: The SF-36 questionnaire, version 2 was a 36-item generic health status measure. SF-36 evaluated 8 health-related aspects of an individual: physical functioning, role-physical, bodily pain, social functioning, mental health, role emotional, vitality, and general health. The score range for each of the 8 health aspects ranged from 0 (worst) to 100 (best), with higher scores indicating good health condition. Two summary scale scores were computed from the 8 health aspect scores: the Physical Component Summary and the Mental Component Summary. Score range for both summary scale ranged from 0 (worst) to 100 (best), with higher scores indicating good health condition.
Time Frame: Baseline, Month 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2233 | 580
units on a scale
  Baseline (n =2233, 580) | 43.51 (11.98) | 43.96 (11.23)
  Month 6 (n =2025, 557) | 48.86 (10.02) | 50.03 (9.14)
  Month 12 (n =1750, 524) | 49.10 (9.89) | 49.78 (9.28)
  Month 24 (n =1362, 442) | 49.22 (9.82) | 49.66 (9.54)
  Month 36 (n =857, 286) | 49.21 (9.95) | 50.17 (8.20)
  Month 48 (n =124, 56) | 50.14 (8.96) | 49.60 (8.24)

75. Secondary Outcome: Number of Participants With Patient Global Assessment (PtGA) Response of "Clear" or "Almost Clear"
Description: The PtGA evaluated the overall skin disease of participants at that point in time on a single-item. Participants provided their response on a 5-point scale ranges from: 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe. Higher score indicated greater severity of disease. Participants who provided their response as "clear (score of 0)" or "almost clear (score of 1)" in PtGA at each specified visit were reported in this outcome measure.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2244 | 583
participants
  Baseline: Clear (n =2244, 583) | 1 | 3
  Baseline: Almost Clear (n =2244, 583) | 25 | 16
  Month 1: Clear (n =2192, 561) | 211 | 127
  Month 1: Almost Clear (n =2192, 561) | 703 | 246
  Month 3: Clear (n =2177, 568) | 248 | 174
  Month 3: Almost Clear (n =2177, 568) | 762 | 254
  Month 6: Clear (n =2030, 562) | 247 | 176
  Month 6: Almost Clear (n =2030, 562) | 748 | 265
  Month 12: Clear (n =1758, 530) | 209 | 151
  Month 12: Almost Clear (n =1758, 530) | 662 | 236
  Month 24: Clear (n =1380, 449) | 171 | 111
  Month 24: Almost Clear (n =1380, 449) | 502 | 202
  Month 36: Clear (n =1112, 377) | 162 | 75
  Month 36: Almost Clear (n =1112, 377) | 418 | 183
  Month 48: Clear (n =410, 125) | 40 | 25
  Month 48: Almost Clear (n =410, 125) | 151 | 60

76. Secondary Outcome: Euro Quality of Life- 5-Dimensions (EQ-5D)-Utility Scores
Description: EQ-5D: participant rated 5-dimension (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) questionnaire to assess health-related quality of life in terms of a single utility score. Each dimension was assessed on a 3-point scale (1=no problems, 2=some problems, 3=extreme problems, where higher scores=worse health condition). The responses from the 5 dimensions were used to calculate a single utility index value. Scoring formula developed by EuroQol Group assigned a utility value for each dimension in the profile. Score was transformed and results in a total score range -0.594 to 1.000; higher score indicated a better health state.
Time Frame: Baseline, Month 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2242 | 581
units on a scale
  Baseline (n =2242, 581) | 0.77 (0.19) | 0.80 (0.17)
  Month 6 (n =2021, 559) | 0.87 (0.15) | 0.91 (0.13)
  Month 12 (n =1750, 523) | 0.88 (0.15) | 0.91 (0.13)
  Month 24 (n =1364, 443) | 0.88 (0.14) | 0.90 (0.14)
  Month 36 (n =857, 284) | 0.88 (0.14) | 0.91 (0.12)
  Month 48 (n =124, 56) | 0.90 (0.13) | 0.89 (0.12)

77. Secondary Outcome: Euro Quality of Life-5-Dimensions (EQ-5D)-Visual Analogue Scale Scores (VAS)
Description: EQ-5D VAS was a participant rated questionnaire to assess health-related quality of life in terms of a single index value. It was a visual analogue scale that ranged from 0 (minimum) to 100 (maximum), with higher scores indicating a better health condition.
Time Frame: Baseline, Month 6, 12, 24, 36, 48
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2224 | 570
units on a scale
  Baseline (n =2224, 570) | 66.39 (23.20) | 68.21 (22.91)
  Month 6 (n =2026, 559) | 78.28 (17.11) | 83.95 (16.18)
  Month 12 (n =1749, 525) | 78.91 (16.95) | 83.80 (14.85)
  Month 24 (n =1365, 443) | 79.80 (16.98) | 83.47 (15.55)
  Month 36 (n =856, 286) | 79.43 (17.01) | 84.62 (14.28)
  Month 48 (n =124, 56) | 82.14 (14.07) | 84.50 (16.87)

78. Secondary Outcome: Number of Participants Who Answered Psoriasis Healthcare Resource Utilization Questionnaire (Ps-HCRU)
Description: Ps-HCRU was a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. In the first section, it assessed direct costs associated with healthcare resource use which included participant's interactions with healthcare providers such as general practitioners, dermatologists, cardiologists, gastroenterologists, psychiatrists, surgeons and nurses. When taking the evening dose of tofacitinib, participants were asked to answer the Ps-HCRU questionnaire only if they had an interaction with a healthcare provider or their work was impacted by psoriasis on that specified day. In this outcome measure, number of participants who answered Ps-HCRU at any specified visits were reported.
Time Frame: Baseline, Month 1, 3, 6, 12, 24, 36, 48
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Number analyzed (Participants) | 2281 | 586
participants
  Baseline | 156 | 44
  Month 1 | 153 | 30
  Month 3 | 204 | 55
  Month 6 | 288 | 71
  Month 12 | 234 | 71
  Month 24 | 171 | 50
  Month 36 | 114 | 30
  Month 48 | 22 | 11

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | Tofacitinib 10 mg | Tofacitinib 5 mg or 10 mg
Serious Adverse Events (participants affected / at risk) | 304/2281 | 88/586
Other Adverse Events (participants affected / at risk) | 1415/2281 | 394/586
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Tofacitinib 10 mg (N=2281) | Tofacitinib 5 mg or 10 mg (N=586)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 3 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1
Atrial flutter (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 5 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 6 | 2
Myocardial ischaemia (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2
Thyroid cyst (Endocrine disorders) | 0 | 1
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 2
Periorbital fat herniation (Eye disorders) | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Salivary gland disorder (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 3 | 0
Fatigue (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 5 | 2
Appendicitis perforated (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 0
Bartonellosis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 6 | 1
Ear infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1
Gastric ulcer helicobacter (Infections and infestations) | 1 | 0
Herpes simplex meningitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 7 | 0
Listeria encephalitis (Infections and infestations) | 1 | 0
Pancreatitis bacterial (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pertussis (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 16 | 5
Pneumonia influenzal (Infections and infestations) | 0 | 2
Post procedural infection (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Purulence (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 1
Viral rash (Infections and infestations) | 1 | 0
Wound abscess (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 3
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 3 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 7 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Wound haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 4 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 2
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm papilla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 4
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Sarcomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Testicular malignant teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hypertonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Calculus urinary (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 4 | 2
Obstructive uropathy (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1/640 | 0/203 — This is gender specific event. The number of participants evaluable for this event are 640 and 203.
Breast pain (Reproductive system and breast disorders) | 0/640 | 1/203 — This is gender specific event. The number of participants evaluable for this event are 640 and 203.
Metrorrhagia (Reproductive system and breast disorders) | 0/640 | 1/203 — This is gender specific event. The number of participants evaluable for this event are 640 and 203.
Ovarian cyst (Reproductive system and breast disorders) | 1/640 | 0/203 — This is gender specific event. The number of participants evaluable for this event are 640 and 203.
Pelvic haematoma (Reproductive system and breast disorders) | 0/640 | 1/203 — This is gender specific event. The number of participants evaluable for this event are 640 and 203.
Prostatism (Reproductive system and breast disorders) | 1/1641 | 0/383 — This is gender specific event. The number of participants evaluable for this event are 1641 and 383.
Uterine polyp (Reproductive system and breast disorders) | 1/640 | 0/203 — This is gender specific event. The number of participants evaluable for this event are 640 and 203.
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 6 | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Severe rebound psoriasis (Investigations) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
Subgaleal haematoma (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 2 | 0
Vein disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 10 mg (N=2281) | Tofacitinib 5 mg or 10 mg (N=586)
Diarrhoea (Gastrointestinal disorders) | 73 | 32
Bronchitis (Infections and infestations) | 134 | 48
Herpes zoster (Infections and infestations) | 136 | 33
Influenza (Infections and infestations) | 126 | 23
Nasopharyngitis (Infections and infestations) | 476 | 122
Upper respiratory tract infection (Infections and infestations) | 264 | 51
Urinary tract infection (Infections and infestations) | 145 | 42
Blood cholesterol increased (Investigations) | 86 | 33
Blood creatine phosphokinase increased (Investigations) | 294 | 92
Gamma-glutamyltransferase increased (Investigations) | 81 | 38
Dyslipidaemia (Metabolism and nutrition disorders) | 73 | 52
Hypercholesterolaemia (Metabolism and nutrition disorders) | 134 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 164 | 40
Headache (Nervous system disorders) | 119 | 38
Psoriasis (Skin and subcutaneous tissue disorders) | 148 | 39
Hypertension (Vascular disorders) | 169 | 44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.